CLINICAL TRIAL: NCT05027438
Title: SEdative-Hypnotic Deprescribing Assisted by a Technology-Driven Insomnia InterVEntion (SEDATIVE)
Brief Title: Reducing Use of Sleep Medications Assisted by a Digital Insomnia Intervention
Acronym: SEDATIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F3732-P; 1I21RX003732-01A1 (NIH)
Record Dates: First submitted 2021-08-20; First posted 2021-08-30 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Insomnia
Keywords: Insomnia; Veterans; Hypnotics and Sedatives; Deprescribing; Cognitive Behavioral Therapy for Insomnia; Telemedicine; Mobile Applications
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Deprescriptions

STUDY DESIGN:
Intervention Model Description: pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COAST + Deprescribing (Experimental): CBT-I with simultaneous sedative-hypnotic deprescribing delivered through a digital platform
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Behavioral: Deprescribing

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — A multimodal psychotherapy that may include stimulus control, sleep restriction, cognitive therapy, psychoeducation, and relaxation strategies
  Other Names: CBT-I
Behavioral: Deprescribing — The reduction or withdrawal of a medication, through gradual dose reduction, managed by a healthcare professional that aims to reduce harm and improve outcomes
  Other Names: Gradual Dose Reduction, Tapering

SUMMARY:
Chronic insomnia is one of the most common health problems among Veterans and significantly impacts their health, function, and quality of life. Sedative-hypnotic medications are the most common treatment despite mixed effectiveness and are associated with numerous risks that can further impact Veteran function. An intervention combining evidence-based interventions for deprescribing sedative-hypnotics and behavioral interventions for insomnia (e.g., Cognitive Behavioral Therapy for Insomnia [CBT-I]) can help to optimize sleep and functional outcomes for Veterans with a desire to reduce or stop using these medications. Furthermore, by delivering these interventions through an easy to use and highly accessible digital platform can provide additional benefits to Veterans, especially those with limited time and access to engage in traditional in-person interventions. The Clinician Operated Assistive Sleep Technology (COAST) is an efficient, scalable, and adaptable platform that can help providers to reach more Veterans and provide evidence-based care that translates to improved health and function.

Aim 1: To assess the feasibility of recruiting Veterans with chronic sedative-hypnotic use to participate in a 12-week combined deprescribing and CBT-I intervention, delivered through the COAST digital platform.

Aim 2: To assess Veteran acceptability and usability of the COAST platform.

Aim 3: To assess change in Veteran sleep, sedative-hypnotic use, and function pre- to post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* A Veteran receiving care at VA Pittsburgh Healthcare System
* Active sedative-hypnotic medication use >14 days/month for >=3 months
* A desire to reduce or stop using sedative-hypnotic medications
* Access to a mobile device with internet

Exclusion Criteria:

* A disorder that would impair participation (e.g., cancer, uncontrolled pain, severe depression)
* A disorder that can be exacerbated by changes in sleep (e.g., seizure disorder, bipolar I disorder)
* High risk of suicide
* An active substance use disorder in past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam D. Bramoweth, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bramoweth AD, Hough CE, McQuillan AD, Spitznogle BL, Thorpe CT, Lickel JJ, Boudreaux-Kelly M, Hamm ME, Germain A. Reduction of Sleep Medications via a Combined Digital Insomnia and Pharmacist-Led Deprescribing Intervention: Protocol for a Feasibility Trial. JMIR Res Protoc. 2023 Jul 20;12:e47636. doi: 10.2196/47636. PMID 37471122

RESULTS

PARTICIPANT FLOW:
Period: Intervention
Arm/Group | COAST + Deprescribing
Started | 36
Completed | 25
Not Completed | 11
Period: Post-Treatment
Arm/Group | COAST + Deprescribing
Started | 25
Completed | 24
Not Completed | 1
Period: 3-month Follow-Up
Arm/Group | COAST + Deprescribing
Started | 24
Completed | 19
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.22 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Marital Status [Count of Participants; unit: Participants]
  Married | 23
  Divorced | 8
  Never Married | 3
  Widowed | 1
  Unknown | 1
Military Branch [Count of Participants; unit: Participants]
  Army | 15
  Marine Corps | 8
  Navy | 6
  Air Force | 5
  Coast Guard | 1
  Unknown | 1
Combat Exposure [Count of Participants; unit: Participants]
  Yes | 21
  No | 15

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI) Change
Description: Total score (0-28): no insomnia (0-7); sub-threshold (8-14); moderate (15-21); and severe insomnia (22-28). A reduction pre- to post-treatment/follow-up of 8 points (or more) indicate a treatment response and a post-treatment/follow-up score or 7 (or less) indicate remission.
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 35
score on a scale
  Baseline | 14.63 (4.04)
  Post-Treatment: number analyzed (Participants) | 24
  Post-Treatment | 6.13 (4.10)
  3-month Follow-Up: number analyzed (Participants) | 18
  3-month Follow-Up | 7.17 (3.59)
Statistical Analysis 1: Comparison: COAST + Deprescribing; baseline to post-treatment; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.58, Standard Deviation 5.19 — post-treatment - baseline (negative value indicates reduction of symptoms); effect size (f2) = 1.42 (large >=0.35)
Statistical Analysis 2: Comparison: COAST + Deprescribing; baseline to 3-month follow-up; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.06, Standard Deviation 4.40 — 3-month follow-up - baseline (negative value indicates reduction of symptoms); effect size (f2) = 1.54 (large >=0.35)

2. Primary Outcome: Sedative-Hypnotic Medication Use Change
Description: Change in dose % from baseline (T0; week 0) to post-treatment (T1; week 12)
  Change in dose % from baseline (T0; week 0) to 3-month follow-up (T2; week 24)
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: % medication dose relative to baseline
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 22
% medication dose relative to baseline
  baseline | 100 (0)
  post-treatment: number analyzed (Participants) | 20
  post-treatment | 41.45 (43.98)
  3-month follow-up | 37.74 (54.93)
Statistical Analysis 1: Comparison: COAST + Deprescribing; % change in medication dose from baseline to post-treatment; Test type: Superiority; p = 0.004, Friedman test — Bonferroni correction; Mean Difference (Net) = 58.55, Standard Deviation 43.98
Statistical Analysis 2: Comparison: COAST + Deprescribing; % change in medication dose from baseline to 3-month follow-up; Test type: Superiority; p = 0.005, Friedman test — Bonferroni correction; Mean Difference (Net) = 62.26, Standard Deviation 54.93

3. Secondary Outcome: Sedative-Hypnotic Medication Cessation
Description: Percentage of participants that stopped using sleep medications at post-treatment (T1; week 12) and 3-month follow-up (T2; week 24)
Time Frame: post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Count of Participants; unit: Participants
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 22
Participants
  post-treatment | 7
  3-month follow-up: number analyzed (Participants) | 20
  3-month follow-up | 12
Statistical Analysis 1: Comparison: COAST + Deprescribing; baseline to post-treatment; Test type: Superiority; p = 0.052, Cochran's Q test; Bonferroni correction; Proportion (%) = 31.8
Statistical Analysis 2: Comparison: COAST + Deprescribing; baseline to 3-month follow-up; Test type: Superiority; p < 0.001, Cochran's Q test; Bonferroni correction; Proportion (%) = 60

4. Secondary Outcome: Sleep Diary - Sleep Onset Latency (SOL) Change
Description: The Sleep Diary measures common sleep variables important for tracking and changing sleep behaviors:
  Sleep Onset Latency (SOL) is the subjective estimate of time it takes to fall asleep after going to bed and turning the lights out (or attempting to go to sleep). SOL is measured in minutes (lower values are better).
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 36
minutes
  baseline | 34.19 (27.73)
  post-treatment: number analyzed (Participants) | 24
  post-treatment | 20.02 (14.50)
  3-month follow-up: number analyzed (Participants) | 22
  3-month follow-up | 20.11 (16.46)
Statistical Analysis 1: Comparison: COAST + Deprescribing; baseline to post-treatment; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -16.67, Standard Deviation 20.57 — post-treatment - baseline (negative value indicates reduction of symptoms); effect size (f2) = 0.54 (large >=0.35)
Statistical Analysis 2: Comparison: COAST + Deprescribing; baseline to 3-month follow-up; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -17.11, Standard Deviation 22.11 — 3-month follow-up - baseline (negative value indicates reduction of symptoms); effect size (f2) = 0.47 (large >=0.35)

5. Secondary Outcome: Sleep Diary - Wake After Sleep Onset (WASO) Change
Description: The Sleep Diary measures common sleep variables important for tracking and changing sleep behaviors:
  Wake After Sleep Onset (WASO) is the subjective estimate of time awake in the middle of the night, after falling asleep and before final rise time/out of bed. WASO is measured in minutes (lower values are better).
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 36
minutes
  baseline | 26.04 (31.90)
  post-treatment: number analyzed (Participants) | 24
  post-treatment | 14.68 (14.96)
  3-month follow-up: number analyzed (Participants) | 22
  3-month follow-up | 11.04 (14.58)
Statistical Analysis 1: Comparison: COAST + Deprescribing; baseline to post-treatment; Test type: Superiority; p = 0.101, Mixed Models Analysis; Mean Difference (Net) = -6.24, Standard Deviation 20.34 — post-treatment - baseline (negative value indicates reduction of symptoms); effect size (f2) = 0.10 (small >=0.02)
Statistical Analysis 2: Comparison: COAST + Deprescribing; baseline to 3-month follow-up; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -10.34, Standard Deviation 18.28 — 3-month follow-up - baseline (negative value indicates reduction of symptoms); effect size (f2) = 0.34 (medium; large >=0.35)

6. Secondary Outcome: Sleep Diary - Sleep Efficiency Change
Description: The Sleep Diary measures common sleep variables important for tracking and changing sleep behaviors:
  Sleep Efficiency (SE) = (total sleep time [TST] / time in bed [TIB]) x 100. SE is measured as a percentage (range 0-100%; higher values are better).
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: sleep efficiency (%)
Arm/Group | COAST + Deprescribing
Number analyzed (Participants) | 36
sleep efficiency (%)
  baseline | 87 (9)
  post-treatment: number analyzed (Participants) | 24
  post-treatment | 93 (5)
  3-month follow-up: number analyzed (Participants) | 22
  3-month follow-up | 94 (5)
Statistical Analysis 1: Comparison: COAST + Deprescribing; baseline to post-treatment; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 5, Standard Deviation 6 — post-treatment - baseline (positive value indicates improvement); effect size (f2) = 0.87 (large >=0.35)
Statistical Analysis 2: Comparison: COAST + Deprescribing; baseline to 3-month follow-up; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 6, Standard Deviation 6 — 3-month follow-up - baseline (positive value indicates improvement); effect size (f2) = 0.96 (large >=0.35)

7. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS 29+2) Change
Description: Includes constructs of Physical Function, Participation in Social Roles, Anxiety, Depression, Fatigue, Sleep Disturbance, Pain Interference and Intensity, and Cognitive Function. Constructs are scored individually (4 items, 4-20) except Cognitive Function (2 items, 2-10).
  T-score: population mean=50 and a standard deviation=10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Anxiety, Depression, Sleep, Pain, and Fatigue, a T-score of 60 is one SD worse than average. By comparison, an Anxiety T-score of 40 is one SD better than average. However, for positively-worded concepts like Physical Function, Cognitive Function, and Social Roles, a T-score of 60 is one SD better than average while a T-score of 40 is one SD worse than average.
  When all constructs are scored together, a preference score is calculated, representing health-related quality of life ranging from 0 (as bad as dead) to 1 (perfect or ideal health).
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- COAST + Deprescribing - Baseline; COAST + Deprescribing - Post-Treatment; COAST + Deprescribing - 3-Month Follow-Up: CBT-I with simultaneous sedative-hypnotic deprescribing delivered through a digital platform
  Cognitive Behavioral Therapy for Insomnia: A multimodal psychotherapy that may include stimulus control, sleep restriction, cognitive therapy, psychoeducation, and relaxation strategies
  Deprescribing: The reduction or withdrawal of a medication, through gradual dose reduction, managed by a healthcare professional that aims to reduce harm and improve outcomes
Arm/Group | COAST + Deprescribing - Baseline | COAST + Deprescribing - Post-Treatment | COAST + Deprescribing - 3-Month Follow-Up
Number analyzed (Participants) | 36 | 24 | 15
T-score
  Anxiety | 51.58 (8.18) | 48.48 (8.51) | 48.39 (7.96)
  Cognitive Function | 45.46 (5.94) | 48.46 (7.60) | 49.98 (4.62)
  Depression | 50.74 (8.77) | 49.08 (8.32) | 46.75 (6.01)
  Fatigue | 56.31 (7.99) | 50.90 (9.17) | 46.93 (8.50)
  Pain Interference/Intensity | 57.74 (6.93) | 56.53 (7.41) | 53.23 (6.38)
  Physical Function | 42.90 (7.30) | 45.40 (6.07) | 47.67 (6.64)
  Sleep Disturbance | 58.48 (6.11) | 50.10 (6.29) | 49.99 (5.22)
  Ability to Participate in Social Roles | 49.07 (8.50) | 54.36 (8.60) | 57.53 (6.63)
Statistical Analysis 1: Comparison: COAST + Deprescribing - Baseline vs COAST + Deprescribing - Post-Treatment; Sleep Disturbance - higher scores indicate more sleep disturbance. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.48, Standard Deviation 6.08 — post-treatment - baseline (negative value indicates improvement); effect size (f2) = 1.14 (large >=0.35)
Statistical Analysis 2: Comparison: COAST + Deprescribing - Baseline vs COAST + Deprescribing - 3-Month Follow-Up; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.82, Standard Deviation 5.62 — 3-month follow-up - baseline (negative value indicates improvement); effect size (f2) = 1.21 (large >=0.35)

8. Secondary Outcome: Patient-Reported Outcomes Measurement Information System Adult Profile (PROMIS 29+2) - PROMIS Preference (PROPr)
Description: The PROMIS-29+2 Profile v2.1 (PROPr) is used to calculate a preference score (PROMIS Preference, PROPr). Preference-based scores provide an overall summary of health-related quality of life on a common metric. Preference-based scores summarize multiple domains on a metric ranging from 0 (as bad as dead) to 1 (perfect or ideal health). Scores can be used in comparisons across groups and for cost-utility analyses. The profile includes all items in the PROMIS-29 Profile v2.1 plus two Cognitive Function Abilities items. T-scores from the measure can be used to calculate a preference-based score.
Time Frame: baseline (T0; week 0), post-treatment (T1; week 12), 3 month follow-up (T2; week 24)
Population: intent to treat analysis - time frame sample size differs due to drop out
Measure: Mean (Standard Deviation); unit: score 0-1
Arm/Group | COAST + Deprescribing - Baseline | COAST + Deprescribing - Post-Treatment | COAST + Deprescribing - 3-Month Follow-Up
Number analyzed (Participants) | 36 | 24 | 14
score 0-1 | 0.29 (0.16) | 0.41 (0.19) | 0.50 (0.15)
Statistical Analysis 1: Comparison: COAST + Deprescribing - Baseline vs COAST + Deprescribing - Post-Treatment; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Net) = 0.11, Standard Deviation 0.21 — post-treatment - baseline (positive value indicates improvement); effect size (f2) = 0.18 (medium >=0.15)
Statistical Analysis 2: Comparison: COAST + Deprescribing - Baseline vs COAST + Deprescribing - 3-Month Follow-Up; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.20, Standard Deviation 0.12 — 3-month follow-up - baseline (positive value indicates improvement); effect size (f2) = 1.99 (large >=0.35)

ADVERSE EVENTS:
Time Frame: Baseline through 3-month follow-up assessment (1 year).
Arm/Group | COAST + Deprescribing
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

LIMITATIONS AND CAVEATS:
Drop out during intervention and failure to complete post-treatment and follow-up assessments resulted in smaller number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT05027438/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT05027438/ICF_000.pdf